CLINICAL TRIAL: NCT00591279
Title: Cancer Control Following Polypectomy
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Mount Sinai Hospital, New York (Other); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); Medical College of Wisconsin (Other); St. Lukes hospital in Racine, Wiscousin (Unknown); Massachusetts General Hospital (Other); Cedars-Sinai Medical Center (Other); Valley Presbyterian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 81-035
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Colon Cancer
Keywords: large bowel cancer; polyps; colorectal cancer
MeSH Terms: conditions — Colonic Neoplasms; Polyps; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fecal occult blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Barium enema and colonoscopy at one and three years after entry.
- B: Barium enema and colonoscopy at three years only after entry.

SUMMARY:
This study evaluates strategies for the surveillance of post-polypectomy patients for the control of bladder cancer

ELIGIBILITY:
Inclusion Criteria:

* referral for colonoscopy or
* referral for proctoscopy or for a complete colonoscopy after a proctoscopy or flexible sigmoidoscopy

Exclusion Criteria:

* prior history of colon cancer, unrelated polypectomy, inflammatory bowel disease, family history of familial polyposis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing colorectal cancer screening
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 1981-02 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
evaluate strategies for the surveillance of post-polypectomy patients | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Sidney Winawer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org